CLINICAL TRIAL: NCT06384521
Title: Type 2 Diabetes Prevention and Management for People With Serious Mental Illness: A Feasibility Study
Brief Title: Lifestyle MIND- Feasibility of Wait-list Control
Acronym: MIND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000500
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes Mellitus; Serious Mental Illness; Schizophrenia; Major Depression; Bipolar Disorder
Keywords: health disparities; integrated care; community engagement
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Schizophrenia; Depressive Disorder, Major; Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Lifestyle MIND
  Interventions: Behavioral: Lifestyle MIND
- Wait-list control arm (Other): Delayed Lifestyle MIND
  Interventions: Behavioral: Lifestyle MIND

INTERVENTIONS:
Behavioral: Lifestyle MIND — Lifestyle MIND is implemented twice a week in the group format, including a physical activities class and a health class. The physical activity class lasts for 60 minutes. Participants engage in physical activities modified from the American College of Sports Medicine guidelines for diabetes. The health class lasts for about 2 hours and is delivered by occupational therapy faculty and students with light refreshments that are friendly for people with diabetes. The first hour of the health class involves psychoeducation and skills training for managing SMI and Type 2 Diabetes Mellitus (T2DM), including topics such as recognizing signs and symptoms of mental disorders and diabetes, goal setting, dealing with setbacks and resistance to change, celebrating culture and holidays, and establishing healthy habits and routines. The second hour of the health class is to address individual needs, social determinants of health, and any needed homework assistance.

SUMMARY:
The goal of this clinical trial is to examine if it is feasible to randomly assign people into two groups and participate in Lifestyle MIND (Mental Illness and/N' Diabetes) at two different times. Lifestyle MIND is a diabetes lifestyle intervention recently developed for people with serious mental illness (SMI). It is known to be helpful for people with SMI who complete it, but the investigators do not know the effect in comparison to those who do not participate in it. The main questions it aims to answer are:

* Does Lifestyle MIND improve diabetes control among people with SMI?
* Will the effect of Lifestyle MIND be sustained 10 weeks after program completion?
* From the provider's perspective, what are the barriers of achieving optimal diabetes treatment outcomes for patients with SMI?

Researchers will compare outcomes of participants in the intervention with those in the wait-list control arm, to see if there will be significant differences in blood glucose level, compliance of diabetes self-management, time staying active, number of emergency department (ED) visits and psychiatric hospitalization, and subjective well-being.

DETAILED DESCRIPTION:
Specific Aims 1 and 2

Study Design:

The study team will do a study called a randomized wait-list control trial. This means the investigators will randomly choose who gets the program first and who waits. Those in the program group will get a 10-week Lifestyle MIND program and then join a self-help group for 10 weeks. The waitlist group will wait for 10 weeks and then get the 10-week Lifestyle MIND program.

Participants:

The study team will recruit 20 people from a program for homeless adults in San Antonio, TX, who often have serious mental illness (SMI). The study team will invite them to an information session to explain the study. After agreeing to join, participants will sign a form and give some basic information after which the study team will randomly assign them to either start the program right away or wait for 10 weeks.

Data Collection and Analysis:

The study team will collect data from all participants at the beginning, after 10 weeks, and after 20 weeks.

Specific Aim 3

To address this aim, the study team will do a qualitative study. Six healthcare professionals, administrators, or leaders who work with people who have both serious mental illness and type 2 diabetes will be interviewed. Questions asked will be:

What works well for helping people with SMI manage their diabetes? What challenges do they face in helping these patients? What could be done to allow them help these patients obtain the best outcomes?

The study team will record and write down the interviews and use a method called thematic analysis to understand the main ideas. We'll use a computer program called NVivo to help us with this.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of SMI
* a diagnosis of T2DM, seeing a health care provider for T2DM, or having been informed by a healthcare provider for being pre-diabetic or diabetic
* willingness to commit to participate for 20 weeks
* ability to respond to self-report scales and questionnaires used in the study

Exclusion Criteria:

* unable to perform the moderate intensity exercise program in Lifestyle MIND

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c) | Weeks 1, 10, and 20
  This is a blood glucose test used to indicate a patient's average blood glucose level in the recent three months. It is a blood glucose measure that's not dominantly affected by the immediate physiological status (e.g., food intakes) at the time of blood drawn. An HbA1c level of 6.5% or higher is diabetic, 5.7 % to 6.4%, prediabetic, and below 5.7%, normal. We will coordinate with the study site and schedule a licensed nurse to take blood samples in designated weeks.
Summary of Diabetes Self-Care Activities (SDSCA) Questionnaire | Weeks 1, 10, and 20
  This is a self-report questionnaire with 11 items to measure a participant's compliance with diabetes self-management including diet, exercise, blood glucose tests, foot care, and smoking status. This questionnaire has been commonly used in diabetes lifestyle intervention studies with good validity and reliability. The Spanish version of this questionnaire is available upon request. Each of the first 10 items is scored on a five-point Likert scale indicating the frequency of the specified behavior as 0 = never to 4 = always. The range of possible scores is 0-40 with a higher score indicating better self management.
Hours of Active and Sedentary Behavior | Weeks 1, 10, and 20
  This is measured by an ActiGraph device which participants will wear on their wrist for a week in Week 1, Week 10, and Week 20. Data of four consecutive days, including the weekend, will be used to calculate the number of hours a participant spends for active and sedentary behaviors. In older adults, the reliability of the ActiGraph measured during daily free-living activities ranged from moderate to excellent (interclass correlation coefficients [ICC]= .75-.89) across intensity categories (i.e., light and moderate intensities) and daily number of steps. In healthy middle-aged adults, the ActiGraph has shown moderate to excellent reliability (ICCs ranged from .74 to .90.
Number of emergency department (ED) visits and psychiatric hospitalizations | Weeks 1, 10, and 20
  ED visits and psychiatric hospitalizations are often the result of poorly managed illness conditions. We will record self-report numbers of ED visits and psychiatric hospitalizations one year before and during the study period.
Satisfaction with Life Scale (SWLS) | Weeks 1, 10, and 20
  This is a 5-item self-report measure of subjective well-being, which is widely used in health research and has good psychometric properties confirmed with the population with SMI. The SWLS total score ranges from 5 to 35, and higher scores indicate better subject well-being. The Spanish translation of SWLS is available upon request.

CONTACTS AND LOCATIONS:
Overall Officials: Chinyu Wu, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No